CLINICAL TRIAL: NCT01103284
Title: A Phase 3, Multinational, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Clinical Efficacy and Safety of DiaPep277 in Newly Diagnosed Type 1 Diabetes Subjects
Brief Title: Efficacy and Safety Study of DiaPep277 in Newly Diagnosed Type 1 Diabetes Adults
Acronym: DIA-AID2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Andromeda Biotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DiaPep277-1001
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: beta-cells; autoimmune; Diabetes; immunomodulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DiaPep277 (Experimental): Administration of 1 mg DiaPep277®, subcutaneously (s.c.) in the upper arm at 0, 1, 3, 6, 9, 12, 15, 18, 21, and 24 months, for a total of 10 administrations.
  Interventions: Drug: DiaPep277
- Placebo (Placebo Comparator): Administration of placebo, subcutaneously (s.c.) in the upper arm at 0, 1, 3, 6, 9, 12, 15, 18, 21, and 24 months, for a total of 10 administrations.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DiaPep277 — 1.0 mg dose in 0.5 mL of solution
  Arms: DiaPep277
Drug: Placebo — 40 mg mannitol in 0.5 mL of solution.
  Dosing: 0, 1, 3, 6, 9, 12, 15, 18, 21, 24 months
  Arms: Placebo

SUMMARY:
This study will look at the treatment effect of DiaPep277 on preservation of beta-cell function, as defined by meal-stimulated secretion of insulin. DiaPep277 is a peptide that changes the way the immune system behaves, stopping its attack on the beta-cells.

Adults (>20 years) with newly diagnosed (<6 months) type 1 diabetes will be treated with 10 injections of DiaPep277 or Placebo over a 2-year treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 1 diabetes within last 6 months
* Age 20-45 years
* fasting basal C-peptide equal or greater than 0.22 nmol/L, lower than 0.8 nmol/L
* BMI between 17 and 30 at screening

Exclusion Criteria:

* Significant disease or condition other than type 1 diabetes
* Diabetes-related complications
* Ongoing treatment with immunosuppressive or immunomodulating agents including chronic corticosteroids

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 475 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah Medical Center, Jerusalem; Thomas Linn, MD, Principal Investigator — University of Giessen; Paolo P Pozzilli, MB, BS, MD, Principal Investigator — University Campus Bio-Medico, Rome; Philip Raskin, MD, Principal Investigator — UT Southwestern Medical Center, Dallas
Locations (75):
- United States (26):
  - Los Gatos, California
  - Sutter Gold Medical Foundation, Modesto, California
  - San Diego Clinical Trials, San Diego, California
  - University of Colorado Hospital - Anschutz Outpatient Pavilion, Aurora, Colorado
  - Creekside Endocrine Associates, Inc., Denver, Colorado
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Innovative Medical Research of South Florida Inc., Aventura, Florida
  - DeLand, Florida
  - Orlando Diabetes & Endocrine Specialists, P.A., Orlando, Florida
  - Tallahassee Endocrine Associates, Tallahassee, Florida
  - Diabetes and Hormonal Disease Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Washington University, St Louis, Missouri
  - Palm Medical Research Center, Las Vegas, Nevada
  - Soutwest Clinical Research Center, LLC, Santa Fe, New Mexico
  - Mountain Diabetes and Endocrine Center, Ashville, North Carolina
  - University of North Carolina Diabetes Care Center, Durham, North Carolina
  - The Lindner Research Center, The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Legacy Clinical Research & Technology Center, Portland, Oregon
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - Cetero Research, San Antonio, Texas
  - Northside Internal Medicine Associates, PS, Spokane, Washington
  - Multicare Specialties Research, Tacoma, Washington
- Austria (2):
  - Universitatsklinik fur Innere Medzin I, Landeskrankenhaus, Innsbruck
  - Rudolfstiftung Hospital, Vienna
- Belarus (5):
  - Endocrinological Unit 1st City Clinical Hospital, Minsk
  - Republican center of Medical Rehabilitation and Balneotherapy, Minsk
  - Health Institution City Endocrinological Dispensary, Minsk
  - Belarusian Medical Academy of Postgraduate Education, Minsk
  - Health Institution Mogilev Diagnostic Center, Mogilev
- Canada (3):
  - LMC Endocrinology Centres, Calgary, Alberta
  - LMC Endocrinology Centres, Oakville, Ontario
  - LMC Endocrinoly Centres, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Kralovske Vinohrady - II. internal department, Prague
  - IKEM/Diabetes Centre/Videnska, Prague
- Tutkimusyksikko, Oulu, Finland
- Germany (5):
  - DDZ Studienzentrum Deutsches Diabetes Zentrum, Düsseldorf
  - Universitatsklinikum Giessen, Giessen
  - Diabetes Centre for Children and Adolescents, Kinderkrankenhaus auf der Bult, Hanover
  - Institut für Diabetesforschung an der Klinik und Hochschulambulanz für Kinder- und Jugendmedizin, München
  - Institut für Diabetesforschung Münster GmbH, Münster
- Hungary (3):
  - University of Szeged Faculty of Medicin, Szeged
  - Veszprem Megyei Csolnoky Ferenc Korhaz es Rendelointezet Diabetologia Centrum, Veszprém
  - Zala Megyei Korhaz es Rendelointezet Diabetologia Centrum, Zalaegerszeg
- Israel (6):
  - Diabetes Clinic Soroka University, Beersheba
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Cent, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Institute for Endocrinology and Diabetes Schneider Children's MC, Petach-Tiqva
- Italy (3):
  - . Endocrinologia e Malattie Metaboliche, Dipartimento biomedico di medicina interna e specialistica, Ex Istituto di clinica medica, Università di Palerm, Palermo
  - Dept. of Endocrinology and Diabetes University Campus Bio-Medico, Rome
  - University La Sapienza, Policlinico Umberto I, Rome
- Lithuania (4):
  - Private Clinic JSC 'Kristavita', Jonava
  - Kaunas Medical University Hospital, Kaunas
  - Public Institution 'Seskines Outpatient Clinic', Vilnius
  - Vilnius Medical University Hospital, Santariskiu Clinic's, Vilnius
- NZOZ OmniMed, Lodz, Poland
- Russia (12):
  - State Educational Institution for Additional Professional Education (SEIAPE) "Ural State Medical, Chelyabinsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Endocrinological scientific center of Rosmedtechnology, Moscow
  - SEIAPE Endocrinology and Diabetology, Moscow
  - City Clinical Hospital #81, Endocrinology Department, Moscow
  - Clinic of New Medical Technology, LLC, Moscow
  - State Healthcare Institution (SHI) "Nizhegorodskaya, Nizhny Novgorod
  - State Healthcare Institution Perm Region Clinical Hospital, Perm
  - St. Petersburg State Healthcare Institution, Saint Petersburg
  - State Educational Institution of Higher Professional Education, Saint Petersburg
  - Limited Liability Company (LLC), Diabetes Center, Samara
  - Siberian State Medical University of Roszdrav, Tomsk
- Spain (2):
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova, Lleida

REFERENCES:
- [Background] Huurman VA, van der Meide PE, Duinkerken G, Willemen S, Cohen IR, Elias D, Roep BO. Immunological efficacy of heat shock protein 60 peptide DiaPep277 therapy in clinical type I diabetes. Clin Exp Immunol. 2008 Jun;152(3):488-97. doi: 10.1111/j.1365-2249.2008.03656.x. Epub 2008 Apr 16. PMID 18422727
- [Background] Huurman VA, Decochez K, Mathieu C, Cohen IR, Roep BO. Therapy with the hsp60 peptide DiaPep277 in C-peptide positive type 1 diabetes patients. Diabetes Metab Res Rev. 2007 May;23(4):269-75. doi: 10.1002/dmrr.691. PMID 17024692
- [Background] Schloot NC, Meierhoff G, Lengyel C, Vandorfi G, Takacs J, Panczel P, Barkai L, Madacsy L, Oroszlan T, Kovacs P, Suto G, Battelino T, Hosszufalusi N, Jermendy G. Effect of heat shock protein peptide DiaPep277 on beta-cell function in paediatric and adult patients with recent-onset diabetes mellitus type 1: two prospective, randomized, double-blind phase II trials. Diabetes Metab Res Rev. 2007 May;23(4):276-85. doi: 10.1002/dmrr.707. PMID 17103487
- [Background] Raz I, Avron A, Tamir M, Metzger M, Symer L, Eldor R, Cohen IR, Elias D. Treatment of new-onset type 1 diabetes with peptide DiaPep277 is safe and associated with preserved beta-cell function: extension of a randomized, double-blind, phase II trial. Diabetes Metab Res Rev. 2007 May;23(4):292-8. doi: 10.1002/dmrr.712. PMID 17124720
- [Background] Eldor R, Kassem S, Raz I. Immune modulation in type 1 diabetes mellitus using DiaPep277: a short review and update of recent clinical trial results. Diabetes Metab Res Rev. 2009 May;25(4):316-20. doi: 10.1002/dmrr.942. PMID 19267355
- [Background] Raz I, Elias D, Avron A, Tamir M, Metzger M, Cohen IR. Beta-cell function in new-onset type 1 diabetes and immunomodulation with a heat-shock protein peptide (DiaPep277): a randomised, double-blind, phase II trial. Lancet. 2001 Nov 24;358(9295):1749-53. doi: 10.1016/S0140-6736(01)06801-5. PMID 11734230
- [Background] Elias D, Avron A, Tamir M, Raz I. DiaPep277 preserves endogenous insulin production by immunomodulation in type 1 diabetes. Ann N Y Acad Sci. 2006 Oct;1079:340-4. doi: 10.1196/annals.1375.052. PMID 17130576
- [Background] Nussbaum G, Zanin-Zhorov A, Quintana F, Lider O, Cohen IR. Peptide p277 of HSP60 signals T cells: inhibition of inflammatory chemotaxis. Int Immunol. 2006 Oct;18(10):1413-9. doi: 10.1093/intimm/dxl074. Epub 2006 Aug 7. PMID 16893923
- [Background] Fischer B, Elias D, Bretzel RG, Linn T. Immunomodulation with heat shock protein DiaPep277 to preserve beta cell function in type 1 diabetes - an update. Expert Opin Biol Ther. 2010 Feb;10(2):265-72. doi: 10.1517/14712590903555176. PMID 20034363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients newly diagnosed with Type 1 diabetes were recruited at medical centers in the US, EU, Argentina, and Israel.
Groups:
- Placebo: Administration of placebo, subcutaneously (s.c.) in the upper arm at 0, 1, 3, 6, 9, 12, 15, 18, 21, and 24 months, for a total of 10 administrations.
  Placebo: 40 mg mannitol in 0.5 mL of solution.
  Dosing: 0, 1, 3, 6, 9, 12, 15, 18, 21, 24 months
Period: Overall Study
Arm/Group | DiaPep277 | Placebo
Started | 236 | 239
Treated | 236 | 238
At Least One Post-baseline Visit (FAS) | 233 (Patients reaching this milestone were included in the Full Analysis Set (FAS) population) | 235 (Patients reaching this milestone were included in the Full Analysis Set (FAS))
Completed | 194 | 195
Not Completed | 42 | 44
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 9 | 10
Not completed — Pregnancy | 3 | 1
Not completed — Protocol Violation | 12 | 5
Not completed — Adverse Event | 0 | 5
Not completed — Withdrawal by Subject | 14 | 18
Not completed — Dermal Hypersensitivity | 0 | 1
Not completed — Termination by the Sponsor | 0 | 1
Not completed — Not described | 2 | 1
Not completed — Missing CRF entries for study completion | 0 | 2

BASELINE CHARACTERISTICS:
Population: All patients randomized into the study are included in presentation of baseline results
Groups:
- Total: Total of all reporting groups
Arm/Group | DiaPep277 | Placebo | Total
Number analyzed (Participants) | 236 | 238 | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.75) | 28.5 (6.56) | 28.6 (6.65)
Age, Customized [Median (Full Range); unit: years] | 27.0 [20 to 45] | 27.0 [20 to 45] | 27.0 [20 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 73 | 152
  Male | 157 | 165 | 322
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 224 | 225 | 449
  Hispanic | 6 | 6 | 12
  Black | 3 | 4 | 7
  Oriental | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Other | 0 | 2 | 2
  Unknown | 1 | 0 | 1
Daily Insulin Dose [Mean (Standard Deviation); unit: IU/kg/day] | 0.305 (0.1587) | 0.317 (0.1649) | 0.311 (0.1618)
Fasting C-Peptide [Mean (Standard Deviation); unit: nmol/L] | 0.388 (0.1473) | 0.407 (0.1731) | 0.398 (0.1609)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucagon-Stimulated C-Peptide AUC at 24 Months
Description: Change in Beta-cell function, measured as stimulated C-peptide secretion 0, 2, 6, 10 and 20 minutes post administration [area under the curve (AUC), 0-20 minutes] at baseline and 24 months, during a glucagon stimulation test (GST). The change in AUC was calculated per patient by subtracting the baseline AUC from the 24 month AUC.
Time Frame: Baseline and 24 months
Population: Full Analysis Set (FAS) All subjects randomized who had a baseline visit and at least one scheduled post-baseline visit
Measure: Mean (Standard Error); unit: nmol*min/L
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 233 | 235
nmol*min/L | -5.20 (0.27) | -4.83 (0.30)
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; The Mixed-Effect Model Repeated Measure (MMRM) was adjusted for the following baseline covariates: age, C-peptide, insulin dose by body weight and AUC

2. Secondary Outcome: Percentage of Subjects That Achieve Good Glycemic Control: HbA1c<7%
Description: The percentage of subjects achieving good glycemic control, i.e. an HbA1c <7% at study end (Month 25). If HbA1c was missing at Month 25, but the Month 24 value was available, then the Month 24 value was used to calculate the percentage of subjects with an HbA1c ≤ 7% at study end.
Time Frame: 24 and 25 months
Population: Full Analysis Set (FAS) All subjects randomized who had a baseline visit and at least one scheduled post-baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 233 | 235
percentage of subjects | 47 [40 to 54] | 47 [40 to 55]
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; Test type: Superiority or Other; p = 0.68, Mixed Models Analysis — A priori threshold for statistical significance was 0.05; The MMRM model was adjusted for the following covariates: age, Baseline C-peptide, Baseline insulin dose adjusted for body weight, and Baseline AUC

3. Other Pre Specified Outcome: Percentage of Subjects Requiring a Daily Insulin Dose ≤ 0.5 IU/kg at End of Study
Description: Percentage of subjects requiring a daily insulin dose ≤ 0.5 IU/kg at end of study (25 Months). If insulin dose was missing at Month 25, but the Month 24 value was available, then the Month 24 value was used to calculate the percentage of subjects with a daily insulin dose ≤ 0.5 IU/kg at study end.
Time Frame: 24 and 25 months
Population: Full Analysis Set (FAS) All subjects randomized who had a baseline visit and at least one scheduled post-baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 233 | 235
percentage of subjects | 63 [57 to 69] | 57 [50 to 63]
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis — The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Frequency of Hypoglycemic Events
Description: Total number of days with at least one hypoglycemic event recorded
Time Frame: Baseline to 25 Months
Population: Full Analysis Set (FAS) All subjects randomized who had a baseline visit and at least one scheduled post-baseline visit
Measure: Number; unit: days
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 233 | 235
days | 1955 | 3264

5. Secondary Outcome: Mean Number of Days With at Least One Hypoglycemic Event
Time Frame: Baseline to 25 months
Population: Full Analysis Set (FAS) All subjects randomized who had a baseline visit and at least one scheduled post-baseline visit
Measure: Mean (Standard Error); unit: days
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 233 | 235
days | 13.0 (2.3) | 35.4 (7.6)
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; The number of hypoglycemia events during the study was analyzed using a negative binomial regression model, with number of events as the dependent variable, and treatment, age, baseline daily insulin dose, and baseline C-peptide as covariates. The log of duration in the study for each patient was used as an offset variable in the model; Test type: Superiority or Other; p = 0.07, negative binomial regression — Standard multiple imputation was used to predict the number and timing of hypoglycemic events after discontinuing the study for subjects who did not remain in the study until Month 25; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [-0.02 to 0.79]

ADVERSE EVENTS:
Time Frame: AE data were collected from the time of subject enrollment through one month after the final product administrations (Total of 25 months after first study product administration)
Arm/Group | DiaPep277 | Placebo
Serious Adverse Events (participants affected / at risk) | 15/236 | 10/238
Other Adverse Events (participants affected / at risk) | 171/236 | 172/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DiaPep277 (N=236) | Placebo (N=238)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0
Tonsillitis Streptococcal (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Meniscus inury (Injury, poisoning and procedural complications) | 1 | 0
multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoglycemic seizure (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DiaPep277 (N=236) | Placebo (N=238)
Nasopharyngitis (Infections and infestations) | 52 | 60
Upper respiratory tract infection (Infections and infestations) | 18 | 13
Influenza (Infections and infestations) | 15 | 17
Sinusitis (Infections and infestations) | 10 | 4
Gastroenteriitis (Infections and infestations) | 7 | 9
Urinary tract infection (Infections and infestations) | 7 | 8
Bronchitis (Infections and infestations) | 7 | 5
Pharyngitis (Infections and infestations) | 5 | 9
Tonsillitis (Infections and infestations) | 4 | 6
Rhinitis (Infections and infestations) | 3 | 9
Nausea (Gastrointestinal disorders) | 9 | 13
Diarrhea (Gastrointestinal disorders) | 9 | 7
Abdominal Pain (Gastrointestinal disorders) | 5 | 6
Toothache (Gastrointestinal disorders) | 5 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4
vomiting (Gastrointestinal disorders) | 4 | 7
Injection site pain (General disorders) | 20 | 18
Asthenia (General disorders) | 3 | 6
Fatigue (General disorders) | 3 | 5
Headache (Nervous system disorders) | 17 | 25
Migraine (Nervous system disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 8
Laceration (Injury, poisoning and procedural complications) | 2 | 5
Joint injury (Injury, poisoning and procedural complications) | 0 | 5
Blood creatine phosphokinase increased (Investigations) | 6 | 3
Blood thyroid stimulating hormone increased (Investigations) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 5
Psychiatric disorders (Psychiatric disorders) | 10 | 9
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 8 | 10
Cardiac disorders (Cardiac disorders) | 8 | 6
Hypothyroidism (Endocrine disorders) | 2 | 5
Immune system disorders (Immune system disorders) | 6 | 6
Hypertension (Vascular disorders) | 2 | 5
Renal and urinary disorders (Renal and urinary disorders) | 4 | 7
Eye disorders (Eye disorders) | 4 | 6
Reproductive system and breast disorders (Reproductive system and breast disorders) | 6 | 4
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall submit any paper or presentation to the Sponsor for review and comments at least 60 days prior to submitting the same to a third party. Upon receiving any request from the Sponsor to delete any Confidential Information or request to delay in publication up to 90 days to allow the filing of any Sponsor application, the Investigator shall take the request action. Investigator shall not be restricted after 18 months from completion of their site's performance in the study.